CLINICAL TRIAL: NCT01569438
Title: A Four-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study Evaluating the Safety and Efficacy of AF-219 in Female Subjects With Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Brief Title: The Safety and Efficacy of Gefapixant (AF-219/MK-7264) in Female Participants With Interstitial Cystitis /Bladder Pain Syndrome (MK-7264-005)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-005; AF219-005 (Other: Afferent Pharmaceuticals); MK-7264-005 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gefapixant (Experimental): Female participants receive gefapixant, a total dose titrated from 50 mg to highest tolerated dose (maximum of 300 mg) twice daily (BID), orally over a period of 6 days with food depending on safety and tolerability, and then maintain that dose for the course of a 4-week treatment period. Participants were allowed to decrease the dose if tolerability issues occurred.
  Interventions: Drug: Gefapixant
- Placebo (Placebo Comparator): Female participants receive dose matched placebo tablets, BID, orally, with food for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — 50 or 300 mg tablets for a total daily dose of 50, 100, 150, 200, 250 or 300 mg BID, orally with food for 4 weeks
  Other Names: AF-219; MK-7264
  Arms: Gefapixant
Drug: Placebo — Dose matched placebo tablets, BID, orally, with food for 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of gefapixant (AF-219/MK-7264) in female participants with moderate to severe pain associated with interstitial cystitis/bladder pain syndrome (IC/BPS) after 4 weeks of treatment.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled, randomized trial designed to assess the efficacy and safety of gefapixant in female participants with moderate to severe pain associated with IC/BPS. The study will consist of 4 phases: Screening, Baseline, Treatment, and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Women of child bearing potential must not be pregnant during the study and must use two forms of birth control
* Clinical evidence of Interstitial Cystitis /Bladder Pain Syndrome (IC/BPS)
* Have provided written informed consent

Exclusion Criteria:

* History of diseases that can be confused for IC/BPS
* Unable to void spontaneously
* Immunosuppressant, intravesicular, nerve stimulator or opioid treatment for certain periods prior to start of the study
* Changes to doses of Elmiron®, antidepressant, alpha-adrenergic antagonist, H1 antagonist, or anti-muscarinic treatment within a certain period prior to the start of the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-04-13 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (40):
- United States (40):
  - Afferent Investigative Site, Glendale, Alabama
  - Afferent Investigative Site, Homewood, Alabama
  - Afferent Investigative Site, Mobile, Alabama
  - Afferent Investigative Site, Phoenix, Arizona
  - Afferent Investigative Site, Glendora, California
  - Afferent Investigative Site, Murrieta, California
  - Afferent Investigative Site, San Diego, California
  - Afferent Investigative Site, Farmington, Connecticut
  - Afferent Investigative Site, New Britain, Connecticut
  - Afferent Investigative Site, Boynton Beach, Florida
  - Afferent Investigative Site, Plantation, Florida
  - Afferent Investigative Site, Coeur d'Alene, Idaho
  - Afferent Investigative Site, Idaho Falls, Idaho
  - Afferent Investigative Site, Meridian, Idaho
  - Afferent Investigative Site, Shreveport, Louisiana
  - Afferent Investigative Site, Annapolis, Maryland
  - Afferent Investigative Site, Ann Arbor, Michigan
  - Afferent Investigative Site, Grand Rapids, Michigan
  - Afferent Investigative Site, Kalamazoo, Michigan
  - Afferent Investigative Site, Royal Oak, Michigan
  - Afferent Investigative Site, Voorhees Township, New Jersey
  - Afferent Investigative Site, Albuquerque, New Mexico
  - Afferent Investigative Site, Brooklyn, New York
  - Afferent Investigative Site, Hyde Park, New York
  - Afferent Investigative Site, Greenville, North Carolina
  - Afferent Investigative Site, Salisbury, North Carolina
  - Afferent Investigative Site, Winston-Salem, North Carolina
  - Afferent Investigative Site, Cincinnati, Ohio
  - Afferent Investigative Site, Cleveland, Ohio
  - Afferent Investigative Site, Tiffin, Ohio
  - Afferent Investigative Site, Zanesville, Ohio
  - Afferent Investigative Site, Bala-Cynwyd, Pennsylvania
  - Afferent Investigative Site, Lancaster, Pennsylvania
  - Afferent Investigative Site, Myrtle Beach, South Carolina
  - Afferent Investigative Site, Dallas, Texas
  - Afferent Investigative Site, Fort Worth, Texas
  - Afferent Investigative Site, Houston, Texas
  - Afferent Investigative Site, Irving, Texas
  - Afferent Investigative Site, Salt Lake City, Utah
  - Afferent Investigative Site, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 107 participants were randomized (55 in Gefapixant intervention group, and 52 in Placebo group).
Pre-assignment Details: Of 107 participants randomized to the study, 105 received at least one dose of study treatment (All Treated Population) and were evaluable for all safety analysis.
Groups:
- Placebo: Female participants receive dose matched placebo tablets, twice daily (BID), orally, with food for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Gefapixant
Started | 52 | 55
Treated | 51 | 54
Titration Set | 38 | 36
Completed | 45 | 33
Not Completed | 7 | 22
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 2 | 15
Not completed — Protocol Violation | 2 | 0
Not completed — Decrease of GFR greater than 30 ml/min | 1 | 0
Not completed — Sponsor/Physician decision | 1 | 1
Not completed — Unable to adhere to study schedule | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant | Placebo | Total
Number analyzed (Participants) | 55 | 52 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 52 | 102
  >=65 years | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 52 | 52 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 46 | 46 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 52 | 107
Numeric Pain Rating Scale (NPRS) Score [Mean (Standard Deviation); unit: Score on a scale] — Participants were instructed to select a number between 0 and 10 where 0 is no pain and 10 is the worst pain possible. The scale was completed by telephone (an interactive voice response system [IVRS]) every evening before bedtime. In order to qualify for study entry, participants must have had an average score of >=4 and <10 during the baseline assessment phase. Population: NPRS score was calculated only on randomized participants who received at least had one dose of study treatment.
  Score on a scale
    number analyzed (Participants) | 54 | 51 | 105
    (all) | 6.20 (1.41) | 6.53 (1.23) | 6.36 (1.33)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Mean Numeric Pain Rating Scale (NPRS) Score at Week 4
Description: The bladder pain severity was measured using 0-10 NPRS, with 0 representing 'no pain' and 10 representing 'the worst pain possible'. Participants were asked to select a number on the scale that best described the severity of bladder pain during past 24 hours over telephone using an interactive voice response system (IVRS) every evening at bedtime during the baseline assessment phase and treatment phase (up to 4 weeks). The primary analysis was conducted using a Mixed Model with Repeated Measures (MMRM) approach to calculate the Least Squares (LS) mean change from baseline in NPRS score and associated Standard Error (SE) at Week 4 for each treatment arm. Negative values indicate decrease in bladder pain severity.
Time Frame: Baseline and Week 4
Population: Titration Completers Population - defined as participants who received at least 1 dose of drug, had at least 1 post-baseline NPRS Score, who titrated the dose in Week 1 of the treatment phase, and who completed the 4-week treatment phase
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 26 | 35
Score on a scale | -2.6 (0.34) | -1.9 (0.31)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; MMRM approach was used to model the change from baseline as a function of treatment, week, treatment by week interaction, baseline score, and baseline score by week interaction; Test type: Other; p = 0.0734, Mixed Model with Repeated Measures — one-sided; Mean Difference = -0.7, 90% CI 2-sided [-1.6 to 0.2]

2. Secondary Outcome: Change From Baseline in Painful Bladder/Interstitial Cystitis Symptom Diary (PBIC-SD) Score at Week 4
Description: To assess the severity of bladder pain syndrome (BPS), an 8-item participant self-report PBIC-SD measure was used. Participants were asked to select a number on the scale that best described the severity of bladder pain over telephone using an IVRS each evening on the three consecutive days (during the Baseline Assessment Phase and during each Treatment Week up to 4 weeks). Each item was graded on a scale from 0 (good condition) to 4 (poor condition) with a total score range 0-32. Higher scores indicate more severe BPS. The analysis was conducted using a MMRM approach to calculate the LS mean change from baseline PBIC-SD total score and associated SE at Week 4 for each treatment arm. Negative values indicate decrease in severity of BPS.
Time Frame: Baseline and Week 4
Population: Titration Completers Population - defined as participants who received at least 1 dose of drug, had at least 1 post-baseline PBIC-SD Score, who titrated the dose in Week 1 of the treatment phase, and who completed the 4-week treatment phase.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 27 | 36
Score on a scale | -7.8 (1.29) | -6.7 (1.15)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2726, Mixed Model With Repeated Measures — one-sided; Mean Difference = -1.0, 90% CI 2-sided [-3.9 to 1.8]

3. Secondary Outcome: Change From Baseline in O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) Score at Week 4
Description: To measure the severity of BPS (urgency and frequency of urination, nighttime urination, and pain or burning) over past month, a 4-item self-report ICSI measure was used. Participants were asked to select a number on the scale that best described the severity of symptoms over telephone using an IVRS every evening at bedtime during the baseline assessment phase and treatment phase (up to 4 weeks). The ICSI score range from 0 (Not at all) to 5 (Almost always) for the first 3 items and a score of 0 (Not at all) to 4 (Almost always) for the last item, with an index score range of 0-19. Higher scores indicate more severe BPS. The analysis was conducted using one-way ANCOVA model to calculate the LS mean change from baseline ICSI total score and associated SE at Week 4 for each treatment arm. Negative values indicate decrease in severity of BPS.
Time Frame: Baseline and Week 4
Population: Titration Completers Population - defined as participants who received at least 1 dose of drug, had at least 1 post-baseline ICSI Score, who titrated the dose in Week 1 of the treatment phase, and who completed the 4-week treatment phase.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 35 | 38
Score on a scale | -3.8 (0.62) | -3.4 (0.60)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; The one-way ANCOVA model was used to calculate change from baseline as a function of treatment and baseline score; Test type: Other; p = 0.3603, ANCOVA — one-sided; Mean Difference = -0.3, 90% CI 2-sided [-1.7 to 1.1]

4. Secondary Outcome: Change From Baseline in Genitourinary Pain Index (GUPI) Score at Week 4
Description: To measure the degree of genitourinary pain symptoms, an 8-item self-report GUPI measure was used. Participants were asked to select a number on the scale that best described the severity of symptoms over telephone using an IVRS every evening at bedtime during the baseline assessment phase and treatment phase (up to 4 weeks). The GUPI instrument yields a total score of 0-45 and 3 subscales: pain (score = 0-23), urinary (score = 0-10), and quality of life (score = 0-12). Higher scores indicate more severe symptoms. The analysis was conducted using one-way ANCOVA model to calculate the LS mean change from baseline GUPI total score and associated SE at Week 4 for each treatment arm. Negative values indicate decrease in degree of genitourinary pain symptoms.
Time Frame: Baseline and Week 4
Population: Titration Completers Population - defined as participants who received at least 1 dose of drug, had at least 1 post-baseline GUPI Score, who titrated the dose in Week 1 of the treatment phase, and who completed the 4-week treatment phase.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 34 | 36
Score on a scale | -5.1 (0.88) | -3.7 (0.86)
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; The one-way ANCOVA model was used to calculate change from baseline as a function of treatment and baseline score; Test type: Other; p = 0.1183, ANCOVA — one-sided; Mean Difference = -1.5, 90% CI 2-sided [-3.5 to 0.6]

ADVERSE EVENTS:
Time Frame: Up to approximately 6 weeks
Description: All-Cause Mortality reported for all randomized participants. Serious Adverse Events (SAEs) and Other Adverse Events (AEs) were reported for all participants who received at least 1 dose of study treatment.
Arm/Group | Placebo | Gefapixant
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/54
Other Adverse Events (participants affected / at risk) | 36/51 | 53/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Gefapixant (N=54)
Dysgeusia (Nervous system disorders) | 9 | 38
Headache (Nervous system disorders) | 6 | 5
Ageusia (Nervous system disorders) | 0 | 7
Hypogeusia (Nervous system disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 10 | 10
Dry mouth (Gastrointestinal disorders) | 2 | 7
Paraesthesia oral (Gastrointestinal disorders) | 0 | 7
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 6
Vomiting (Gastrointestinal disorders) | 1 | 5
Hypoaesthesia oral (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Pollakiuria (Renal and urinary disorders) | 3 | 5
Dysuria (Renal and urinary disorders) | 1 | 4
Bladder pain (Renal and urinary disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Urine output decreased (Investigations) | 1 | 7
Urinary tract infection (Infections and infestations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
60 days prior to the submission of any results, the PI shall submit to SPONSOR any proposed PUBLICATION, which period may be extended for an additional 30 days if requested by SPONSOR. If any Confidential Information should be redacted or patent applications relating to an Invention should be filed prior to PUBLICATION, then PUBLICATION will be delayed until patent application has been filed. Delay of a PUBLICATION shall not exceed 24 months from the date of such notice to the PI.